CLINICAL TRIAL: NCT03723226
Title: Impact of Low-Intensity Resistance Exercise With and Without Blood Flow Redistricted (BFR) on Muscle Mitochondrial Oxidative Capacity
Brief Title: BFR and Muscle Mitochondrial Oxidative Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University and A&M College (Other)
Collaborators: Delfi, Inc. (Unknown)
Responsible Party: Principal Investigator, Brian Irving, Assistant Professor, Louisiana State University and A&M College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB#3934
Record Dates: First submitted 2018-09-21; First posted 2018-10-29 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Mitochondria; Strength; Hypertrophy
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Load Resistance Exercise (Active Comparator): Subjects allocated to Low Load Resistance Exercise will undergo 6 weeks of single-legged low load (25%) resistance exercise. Their contralateral leg will serve as within subject control.
  Interventions: Behavioral: Low Load Resistance Exercise
- Low Load Resistance Exercise + BFR (Experimental): Subjects allocated to Low Load Resistance Exercise + BFR will undergo 6 weeks of single-legged low load (25%) resistance exercise plus blood flow restriction. Their contralateral leg will serve as within subject control.
  Interventions: Behavioral: Low Load Resistance Exercise + BFR

INTERVENTIONS:
Behavioral: Low Load Resistance Exercise — Subjects allocated to Low Load Resistance Exercise will undergo 6 weeks of single-legged low load (25%) resistance exercise. Subjects will then perform 4 sets of 30, 15, 15 and 15 repetitions at 25% of their 1RM for the single-legged leg press and single-legged knee extensions. Their contralateral leg will serve as within subject control.
  Arms: Low Load Resistance Exercise
Behavioral: Low Load Resistance Exercise + BFR — Subjects allocated to Low Load Resistance Exercise + BFR will undergo 6 weeks of single-legged low load (25%) resistance exercise with blood flow restriction (60% occlusion pressure). Subjects will then perform 4 sets of 30, 15, 15 and 15 repetitions at 25% of their 1RM for the single-legged leg press and single-legged knee extensions. Their contralateral leg will serve as within subject control.
  Arms: Low Load Resistance Exercise + BFR

SUMMARY:
Blood flow restricted (BFR) exercise has been shown to improve skeletal muscle adaptations to resistance exercise. BFR uses blood pressure cuffs (i.e., tourniquets) to reduce skeletal muscle blood flow during resistance exercise. One benefit of BFR is that skeletal muscle adaptations to resistance exercise training including muscle hypertrophy and increases in strength can be achieved at lower-loads (e.g., 25-30% 1RM), that are often comparable to more traditional resistance training loads (70-85% 1RM). However, the impact that low-load BFR resistance exercise has on muscle quality and bioenergetics is unknown. The present study will examine the impact of 6 weeks of low-load, single-leg resistance exercise training with or without personalized BFR on measures of muscle mass, strength, quality, and mitochondrial bioenergetics. The investigators will recruit and study up to 30, previously sedentary, healthy, college-aged adults (18-40 years). The investigators will measure muscle mass using Dual Energy X-Ray Absorptiometry and muscle strength and endurance using isokinetic testing. The investigators will normalize knee extensor strength to lower limb lean mass to quantify muscle quality. The investigators will also use near infrared spectroscopy (NIRS) to measure mitochondrial oxidative capacity in the vastus lateralis. Finally, the investigators will measure markers of systemic inflammation and markers of muscle damage using commercially available ELISA assays.

ELIGIBILITY:
Inclusion Criteria.

1. Capable and willing to give written informed consent
2. Capable of understanding inclusion and exclusion criteria
3. 18-40 years of age inclusive
4. Body Mass Index (BMI) between 18.5-30 kg/m2 inclusive
5. No medical condition that would limit their participation in supervised exercise training based on the Physical Activity Readiness Questionnaire for Everyone (PARQ+)
6. No current prescription medications, with the exception of birth control
7. Willing to allow researchers to use data, biospecimens (e.g., blood) and images (e.g., Dual Energy x-Ray Absorptiometry) for research purposes after study participation is completed

Exclusion Criteria.

1. Evidence or self-report being pregnant, lactating, or anticipating becoming pregnant in the next year
2. Participation in resistance or aerobic exercise training > 2 days per week within the 3 months prior to screening
3. Self-report of history of type 1 or 2 diabetes mellitus
4. Self-report history of cardiovascular, peripheral vascular, cerebral vascular, pulmonary, or renal disease
5. Self-report or evidence of uncontrolled hypertension
6. Self-report history of blood clotting disorders
7. Self-report history of deep vein thrombosis or pulmonary embolism
8. Self-report history of sickle cell trait
9. Self-report history of varicose veins
10. Self-report history of a myopathy leading to muscle loss, weakness, severe cramps or myalgia
11. Self-report history of orthopedic limitations that would preclude them from participation in a dynamic exercise program
12. Self-report history of musculoskeletal disorders (e.g., severe osteoarthritis, rheumatoid arthritis, avascular necrosis or osteonecrosis)
13. Self-report history of neurological disorders (e.g., peripheral neuropathy, amyotrophic lateral sclerosis, multiple sclerosis, fibromyalgia, Parkinson's disease)
14. Weight loss of > 10% in the last 3 months prior to screening
15. Active smoking
16. Current consumption of > 14 alcoholic drinks per week based on self-report
17. Absolute Contraindication to Exercise as Defined by the American College of Sports Medicine,1 including:

    1. Resting diastolic blood pressure > 100 mm Hg
    2. Resting systolic blood pressure > 180 mm Hg
    3. Resting heart rate > 100 beats per min
18. Self-report acute viral or bacterial upper or lower respiratory infection at screening
19. Any other condition that in the judgement of the Principal Investigator and/or the Medical Director of this protocol may interfere with study participation and adherence to the protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in Mitochondrial Oxidative Capacity | Changes from baseline (pre-training) to follow-up (about 48-72 hours post-training).
  Changes in mitochondrial oxidative capacity will be measured using near infrared spectroscopy (NIRS).

SECONDARY OUTCOMES:
Changes in Muscle Mass measured by Dual Energy X-ray Absorptiometry | Changes from baseline (pre-training) to follow-up (about 48-72 hours post-training)
  Changes in muscle mass will be measured by Dual Energy X-ray Absorptiometry
Changes in Muscle Strength measured using Isokinetic Dynamometry | Changes from baseline (pre-training) to follow-up (about 48-72 hours post-training)
  Changes in muscle strength measured using isokinetic dynamometry
Changes in Muscle Endurance measured using Isokinetic Dynamometry | Changes from baseline (pre-training) to follow-up (about 48-72 hours post-training)
  Changes in muscle endurance measured using isokinetic dynamometry

CONTACTS AND LOCATIONS:
Overall Officials: Brian Irving, PhD, Principal Investigator — Louisiana State University - Kinesiology
Locations (1):
- Lousiana State University, Baton Rouge, Louisiana, United States